CLINICAL TRIAL: NCT06690411
Title: Effectiveness of Myofascial Release and Mulligan Concept Techniques in Patients With Cervicogenic Headache: A Single Blind-Randomized Clinical Trial
Brief Title: Comparison of Myofascial Release and Mulligan Concept Techniques in Patients With Cervicogenic Headache
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Istanbul Kent University (Other)
Responsible Party: Principal Investigator, fatih bali, Lecturer, Assoc. Dr., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-4329
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cervicogenic Headache; Cervicogenic Headaches
Keywords: Cervicogenic headache; Mulligan SNAG; Myofascial Release; Physiotherapy; Headache; Manual Therapy
MeSH Terms: conditions — Post-Traumatic Headache; Headache | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: This study will be a single blind-randomized clinical trial. The researcher who makes the evaluations will not know which treatment the individuals received, in other words, will be blind to the groups.
Who Masked: Outcomes Assessor
Masking Description: The researcher who makes the evaluations will not know which treatment the individuals received, in other words, will be blind to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release Group (Experimental): Twenty participants who will be randomized into the myofascial release group will undergo the myofascial release technique by an experienced physiotherapist 3 times a week for 4 weeks.
  Interventions: Other: Myofascial Release Technique
- Mulligan SNAG group (Experimental): Twenty participants who will be randomized into the Mulligan SNAG group will undergo the Mulligan SNAG technique by an experienced physiotherapist 3 times a week for 4 weeks.
  Interventions: Other: Mulligan Concept

INTERVENTIONS:
Other: Mulligan Concept — The participants of the Mulligan SNAG group will undergo the Mulligan SNAG technique. Mulligan's SNAG technique is a gentle manual therapy method. This technique is based on the correction of the joint position. There are 3 techniques specified for headache; Headache SNAG, Reverse Headache SNAG, and C1-C2 SNAG.
  Arms: Mulligan SNAG group
Other: Myofascial Release Technique — Myofascial therapy can be described as massage-type manual therapy. The participants of the Myofascial Release Group will undergo the myofascial release technique.
  Arms: Myofascial Release Group

SUMMARY:
The International Headache Society classifies cervicogenic headache as a secondary headache caused by a disorder of the cervical spine and its components. Mulligan Concept (SNAG) is a gentle manual therapy that can be applied to the neck area. The myofascial release technique is also a massage-type manual therapy technique that is widely used in physiotherapy to relieve pain and tension in the relevant muscle group.

This clinical trial aims to investigate the effectiveness of the Mulligan Concept and myofascial release technique in patients with cervicogenic headaches. The main questions it aims to answer are:

1. Does the Mulligan Concept improve hand grip strength, pressure pain threshold, range of motion, pain frequency, pain intensity, pain duration, number of medications used, daily living activities, and disability in patients with cervicogenic headache?
2. Does myofascial release technique improve hand grip strength, pressure pain threshold, range of motion, pain frequency, pain intensity, pain duration, number of medications used, daily living activities, and disability in patients with cervicogenic headache?

Researchers will compare the Mulligan Concept to a myofascial release technique to see which physiotherapy method has more significant results in treating cervicogenic headaches.

Participants will:

* Undergo the evaluations mentioned above before and after interventions
* Undergo Mulligan Concept applications or the myofascial release technique 3 times a week for 4 weeks
* Keep a diary of their symptoms and the number of times they use a drug

DETAILED DESCRIPTION:
Although headache is one of the most common neurological symptoms, it is still not fully recognized and treated worldwide. The International Headache Society divides headaches into primary and secondary categories. The International Headache Society classifies cervicogenic headache as a secondary headache caused by a disorder of the cervical spine and its components. The prevalence in the general population is estimated to be approximately 0.17% to 4.1%.

Cervicogenic headache features are as follows;

1. observed in adulthood,
2. unilateral and does not change sides,
3. radiating from the back of the head and neck to the ear and cheekbone,
4. can be triggered mechanically by maneuvers,
5. characterized by compressive pain that starts seconds or 30 minutes after the maneuver and lasts for several days to weeks

The diagnostic criteria for cervicogenic headache are as follows:

1. The headache developed at a time similar to the onset of the cervical disorder or the appearance of the lesion
2. The headache has significantly decreased or disappeared in parallel with the regression or complete healing of the cervical disorder or lesion
3. The cervical range of motion is reduced and the headache worsens significantly with stimulating maneuvers
4. The headache disappears after the cervical structure or nerve source is blocked for diagnosis

Studies show that physiotherapy and rehabilitation approaches such as manual therapy, exercise training, and dry needling are effective in treating headaches.

Studies have shown that people with cervicogenic headaches have a high rate of C1-C2 dysfunction. The mechanism of Mulligan's movement mobilization technique (SNAG) is based on the correction of joint position. Mulligan's SNAG technique is a gentle manual therapy method. Some studies have shown that Mulligan mobilization increases the range of motion and significantly reduces pain intensity and frequency in patients with cervicogenic headaches

Another form of massage-type manual therapy, myofascial release, is widely used in clinical practice. Previous studies have found that active myofascial trigger points often trigger tension-type headaches and migraines with palpation. Therefore, treatment of these myofascial trigger points may be an effective headache management.

In light of the literature data, this study aims to investigate and compare the effectiveness of physiotherapy methods such as Mulligan Concept applications and myofascial release technique on hand grip strength, pressure pain threshold, range of motion, pain frequency, pain intensity, pain duration, number of medication use, daily living activities and disability in patients with cervicogenic headache.

Hypotheses of this study are;

H0: There is no significant difference in favor of myofascial release technique or Mulligan concept applications in terms of pressure pain threshold, neck joint range of motion, handgrip strength, pain intensity, frequency and duration, number of medications used, disability and daily living activities between myofascial release technique and Mulligan concept applications in cervicogenic headache.

H1: There is a significant difference in favor of myofascial release technique between myofascial release technique and Mulligan concept applications in terms of pressure pain threshold, neck joint range of motion, handgrip strength, pain intensity, frequency and duration, number of medications used, disability and daily living activities between myofascial release technique and Mulligan concept applications in cervicogenic headache.

H2: There is a significant difference in favor of Mulligan concept applications between myofascial release technique and Mulligan concept applications in terms of pressure pain threshold, neck joint range of motion, handgrip strength, pain intensity, frequency and duration, number of medications used, disability and daily living activities.

To determine whether the physiotherapy approach produces greater significant outcomes for treating cervicogenic headaches, researchers will compare the Mulligan Concept with a myofascial release technique.

The 40 individuals, consisting of women and men, who will participate in the study will be randomly divided into two groups. These groups will consist of individuals who receive the myofascial release method or the Mulligan concept technique. After the initial evaluations, both groups will be applied to a 4-week treatment program consisting of 3 sessions per week and the evaluations will be repeated at the end of the 4 weeks. The researcher who makes the evaluations will not know which treatment the individuals received, in other words, will be blind to the groups.

The participants will be evaluated on their neck joint range of motion, pressure pain threshold, hand grip strength, headache and functionality, and disability due to neck problems. In addition, they will be evaluated on their pain frequency, intensity, and duration. Participants will keep a diary of their symptoms and the number of times they use a medication.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with cervicogenic headache according to the International Classification of Headache Disorder-III diagnostic criteria
* Having been diagnosed with cervicogenic headache for more than 3 months
* Having a headache accompanying neck pain
* Having restricted neck joint movement according to the Flexion-Rotation Test
* Having pain between 3 and 8 according to the Visual Analog Scale
* Being between 25-60 years of age
* Agreeing to participate in the study voluntarily

Exclusion Criteria:

* Previous cervical surgery
* Previous cervical trauma
* Having received diagnosis-related physiotherapy in the last 6 months
* Diagnosis of tumor or cancer
* Having other types of headache
* Serious cardiovascular, cerebrovascular, hematological, metabolic, neurological or mental disease
* Being pregnant or breastfeeding
* Having red flags for manual therapy
* Dizziness with headache, visual disturbance
* Congenital cervical disorder
* Rheumatoid arthritis, cervical spondylolisthesis, cervical instability, infection

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Test-6 | 10 minutes
  Headache Impact Test-6 (HIT-6) evaluates the effects of headaches on daily living activities. HIT-6 shows good internal consistency, retest reliability, validity and responsiveness. A total score of 36 is the best in terms of headache, and 78 is the worst. In this study, HIT-6 will be used to evaluate how headache affects individuals' daily living activities.
Hand Grip Strength Measurement | 1 minute
  To the best of our knowledge, no previous study has evaluated the effect of headache on handgrip strength. However, studies have shown a negative correlation between neck pain and handgrip strength. The Jamar Hand Dynamometer is the gold standard tool for handgrip strength assessment in clinical and research settings with its validity and reliability. In this study, Jamar dynamometer will be used to evaluate the hand grip strength of patients on the affected side.

SECONDARY OUTCOMES:
Muscle Tone Measurement | 5 minutes
  In this study, MyotonPro will be used to evaluate the effect of physiotherapy techniques on muscle tone. MyotonPRO offers a non-invasive, reliable and accurate solution for digital palpation of soft biological tissues. The device measures superficial skeletal muscles, tendons, ligaments, adipose tissue and skin. MyotonPRO is a hand-held, smartphone-sized device which is quick and easy to use. Scientific research has proven its practicality and versatility.
Cervical Range of Motion Measurement | 5 minutes
  A reduction in the cervical joint range of motion is frequently observed in cervicogenic headaches. A digital goniometer is a valid and reliable tool for measuring joint range of motion in individuals. In this study, digital goniometer; C1-C2 Flexion-Rotation Test will be used to evaluate flexion-extension, right and left rotation neck joint range of motion.
Pain Pressure Threshold Measurement | 5 minutes
  Pain pressure threshold measurement will be performed to assess pain sensitivity and determine pressure perception. The algometer is the gold standard tool for pain pressure threshold measurement. In this study, pressure pain threshold assessment will be performed on the trapezius muscle and suboccipital muscles on the affected side of the patients.
Neck Disability Index | 10 minutes
  Neck Disability Index is a ten-part test that determines how neck pain affects daily living activities. The Neck Disability Index is a self-scored disability instrument used in patients with cervical musculoskeletal disorders but is increasingly being used to assess neck pain-related disability in individuals with headaches. In this study, NDI will be used to evaluate how patients' neck problems affect their daily living activities. The minimum score is 0, maximum score is 100. High scores show worse results, while low scores show better results.
Diary | 3 minutes a day
  The diary helps both users and healthcare professionals assess the impact of headaches, make diagnoses, and inform healthcare decision-making. In this study, a headache diary will be used to assess patients' headache intensity, frequency, duration, and medication use.
Postural Examination | 3 minutes
  Anterior translations of the head or shoulder may contribute to pain in the upper half of the body. In this study, head and neck translations will be evaluated by measuring the wall-tragus distance and the craniovertebral angle (C7-tragus horizontal angle). Optimal angle of the craniovertebral angle is 48-50.

CONTACTS AND LOCATIONS:
Locations (1):
- Sefakoy Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Correll S, Field J, Hutchinson H, Mickevicius G, Fitzsimmons A, Smoot B. RELIABILITY AND VALIDITY OF THE HALO DIGITAL GONIOMETER FOR SHOULDER RANGE OF MOTION IN HEALTHY SUBJECTS. Int J Sports Phys Ther. 2018 Aug;13(4):707-714. PMID 30140564
- [Background] Corum M, Aydin T, Medin Ceylan C, Kesiktas FN. The comparative effects of spinal manipulation, myofascial release and exercise in tension-type headache patients with neck pain: A randomized controlled trial. Complement Ther Clin Pract. 2021 May;43:101319. doi: 10.1016/j.ctcp.2021.101319. Epub 2021 Jan 24. PMID 33517104
- [Background] Liang Z, Thomas L, Jull G, Treleaven J. The Neck Disability Index Reflects Allodynia and Headache Disability but Not Cervical Musculoskeletal Dysfunction in Migraine. Phys Ther. 2022 May 5;102(5):pzac027. doi: 10.1093/ptj/pzac027. PMID 35230421